CLINICAL TRIAL: NCT03387228
Title: Pain Education for Patients With Non-specific Low Back Pain in Nepal: A Feasibility Clinical Trial
Brief Title: Pain Education for Patients With Low Back Pain in Nepal: A Feasibility Study
Acronym: PEN-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Collaborators: University of Otago (Other); University of Washington (Other); University of South Australia (Other)
Responsible Party: Principal Investigator, Saurab Sharma, Assistant Professor, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NHRC-422/2017
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Low Back Pain, Mechanical
Keywords: back pain; low back pain; Explain Pain; Pain education
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Feasibility of a two group randomized clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor and statistician performing data analysis will be masked for the group allocation of all the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain education group (PEG) (Experimental): Pain education based on Explain Pain developed by Moseley and Butler in 2003.
  Interventions: Other: Pain education
- Control group (CG) (Active Comparator): Evidence based physiotherapy care brief education, superficial heat, massage, and exercise.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Pain education — Pain education intervention we plan to use is based on Explain Pain developed by Moseley and Butler in 2003. The pain education handout and materials produced in Nepali will be proof-read and pre-tested in 5 - 10 Nepalese with LBP as needed, and corrected, if necessary.
  Dosage: A single (approximately) one hour pain education will be delivered to the PEG.
  Home advice: A printed handout of the pain education material will be provided only to the study participants in the PEG. Participants will be advised to read them (or have family members read them), followed by walking for 30 minutes.
  Arms: Pain education group (PEG)
Other: Control group — The control participants will receive physiotherapy care based on the recent clinical practice guidelines. This control group intervention will comprise of: (1) education (advice to remain active); (2) massage to back; (3) superficial heat; and (4) static cycling or (treadmill) walking with the aim to promote physical activity. Although superficial heat is recommended in the acute/subacute LBP, we included this as a common treatment for all types of LBP including chronic LBP, which could be a part of self-management.
  Duration of treatment: 1 hour. Home advice: Participants will be advised to self-manage their back pain based on the information provided. Home exercise leaflet with emphasis on the value of exercise to increase strength and endurance, followed by a 30 minutes walking.
  Arms: Control group (CG)

SUMMARY:
The primary aim of this study is to evaluate the feasibility of a full randomized clinical trial for assessing the effects of pain education as an intervention for patients with LBP in a physiotherapy facility in Nepal. The primary objectives of the study are related to feasibility of randomized clinical trial including: (1) willingness to participate in a clinical trial, (2) acceptability of random allocation to one of the two study groups, (3) feasibility of blinding the assessor(s), (4) eligibility and recruitment rates, (5) acceptability of screening procedures, (6) possible contamination between the groups, (7) credibility of pain education for patients with LBP, (8) adherence to intervention, (9) satisfaction of treatment, and (10) difficulty in understanding the content of pain education.

To address the study objectives, an assessor-blinded, two arm randomized feasibility study was designed. Forty patients with LBP will be randomly allocated to one of the two study arms, (1) pain education in the experimental group, and (2) evidence based care in the control group (CG).

DETAILED DESCRIPTION:
This is a feasibility study that is being performed to determine if a full randomized controlled trial (RCT) can be successfully conducted and if it should be conducted. The definition of a feasibility study highlights the question, "Can this study be done?" The SPIRIT statement and the CONSORT statement- extension to pilot and feasibility randomized study will be followed in the planning and reporting of the protocol and the manuscript of this feasibility study respectively.

The study will be assessor blind two-arm feasibility clinical trial study. Ethical approval was obtained from the Nepal Health Research Council (NHRC) and University of Otago Human Ethics Committee. The study will be conducted in the Sahara Rehabilitation Hospital, Kathmandu, Nepal which is a private hospital in Kathmandu, Nepal.

Overview of the study: Advertisement of the study will be made in social media. Interested candidates will be screened for eligibility. Eligible patients with LBP will be enrolled in the study. Participants will be randomly assigned to one of the two groups. All the participants in the experimental group will receive pain education and those in the control group will receive usual (evidence based) physiotherapy care. All the participants will be assessed at baseline, and follow-up assessment approximately after a week of randomization.

Participant screening and recruitment: Consecutive participants with non-specific low back pain will be invited to participate in this study. Interested candidates will be explained the study purpose, benefits and harms of the intervention, time required for the completion of the study, follow-up duration, voluntary nature of participation, cost of participation, and the rights to withdraw from the study at any point. A participant information sheet will be provided to all potential participants. If the potential participants are interested in participating, they will be screened for eligibility by a research assistant who is a physiotherapist. If the participants are found eligible, informed consent will be obtained. For those who cannot sign the consent, a witness will sign on their behalf, or the study participant will provide a thumb print on the form for those who cannot write or sign the form as per the ethical guidelines provided by NHRC. Patients with no education and who cannot sign an informed consent will be included in order to increase the inclusion of uneducated or low education group, given that 31% people in Nepal who are five years old or more cannot read and write. Additionally, exploration of feasibility of pain education in those with no schooling or low educational attainment is important in order to inform clinical practice.

Participants will be informed that they will receive one of the two treatments randomly. It will be highlighted that both of the treatment options are thought to be effective for low back pain, and that the goal of the main study is to compare the interventions, however the current study will more specifically evaluate the feasibility of such a study. There will be no restriction on the participants on both the groups in the pharmacological interventions they receive, however, participants in the intervention group will be restricted on receiving other physiotherapy interventions on day 1 only. All the participants will continue to receive the regular interventions provided by the centre from the second visit after follow-up assessment in the second week.

Group Allocation, Randomization and Blinding: Random number sequence will be generated by a researcher not involved in data collection or providing treatment using www.random.org. Allocation concealment will be performed using opaque, sealed envelopes. The participants will be allocated to one of the two groups by a hospital staff who is not the assessor. The two groups are: Group 1: Pain education group (PEG); and Group 2: Control group (CG).

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific LBP (LBP other than those excluded, see exclusion criteria below),
* any duration with pain,
* pain primarily localized between T12 and gluteal folds,
* age 18 years or older,
* average pain intensity reported as moderate, or severe, or very severe on a PROMIS five- point PROMIS Pain Intensity Short-form Scale over the past week,
* is a Nepalese and is able to understand and speak Nepali fluently.

Exclusion Criteria:

* Participants with likely specific causes of LBP will be excluded using a triage procedure as suggested by Bardin and colleagues,
* having history of prolonged use of corticosteroid,
* history of malignancy,
* recent history of fever or chills,
* history of other diseases associated with compromise in immune system,
* history of recent spinal surgery or dental procedures,
* history of recent history of trauma to spine or a spine fracture,
* history of bladder and bowel dysfunction,
* history of perineal or saddle anaesthesia,
* history of weakness of lower extremity or loss of sensation in lower extremity. -
* current pregnancy,
* history of diagnosed mental health conditions (e.g., schizophrenia, bipolar disorder, major depressive disorder) that would limit successful participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment 1: Willingness to participate in a clinical trial | During the enrollment
  All the consecutive participants presenting at the physiotherapy department will be explained about the study and invited to participate in the study. The number of participants not willing to participate will be recorded with the reason for not wanting to participate. Total number of patients not willing to participate will be recorded with the reasons not to participate.
Feasibility of recruitment 2: Eligibility and recruitment | During the enrollment
  The total number of participants screened, found eligible, and recruited will be recorded during the screening and recruitment process. The reasons why the participants were ineligible for inclusion in the study will be recorded for every participant who did not meet the eligibility criteria. If the participants refused to participate in the study, the reasons for refusal will be recorded. Finally, the consent rates will be recorded. The number of participants screened, who were eligible, who consented to participate, who refused to participate, reasons for exclusion and refusal will be reported as frequencies.
Feasibility of blinding the assessor | Final assessment at 1 week follow up
  By asking the assessor two questions at the end of the follow-up assessment: (1) Did you receive any information that indicated which group the participant belonged to? and (2) How did you receive information about which group the patients belonged to? Assessor's guess if the participants belonged to experimental or control group will be recorded. The responses will be coded as 'correct guess' or 'incorrect guess.' The frequency of "yes" and "no" as the answer to the first question will be counted. The frequency of the correct and incorrect guesses will also be counted. Finally, reasons for guesses will qualitatively analyzed.
Acceptability of screening procedures and random allocation | During the enrollment
  The lead researcher will interview the physiotherapist(s) screening the patients for eligibility by asking the following open-ended question at the end of every week, "Were there any difficulties or challenges in screening and recruiting the participants the past week?" The responses will be recorded as 'Yes' or 'No'.
  The assessor will ask all the participants during recruitment if randomly allocating one of the two treatments is acceptable to them.
Understanding possible contamination between the groups | Final assessment at 1 week
  Contamination between the groups will be assessed by asking all the participant of the study the following questions at the follow-up assessment: (1) "Have you talked to other participants in this study about the intervention they are receiving?"; If yes, further ask, "Was your attitude towards the intervention, or intervention changed after talking to one of the participants in the other group?"; (2) "Are you aware of the intervention that any participants in the other group are receiving in the study?"; and (3) Are any of the participants in the other group aware of the type of intervention you are receiving in this study?" Participants in the usual care group will be asked the following question: "Did you read the pain education booklet or watch the video which is one of the components of the intervention group?"
Credibility and acceptability of the interventions | Baseline assessment and follow up 1 week assessment
  It will be assessed using five questions. Responses for each of the five questions will be recorded on a Likert Scale where, 0= "Not at all", 1= "A little bit", 2= "Somewhat", 3= "Quite a bit", 4= "Very much."
Adherence to the intervention | Baseline assessment and final assessment at 1 week
  Adherence to home treatment will be assessed by asking the participants in both groups to maintain a log of home treatment, in which the participants will tick mark a box for every day for a total of five days. Total number of responses will be computed by adding the number of days. Adherence will be computed by summing total number of home interventions in each group, represented by a discrete number. Reasons for non-adherence will be listed and analyzed qualitatively.
Satisfaction of treatment | Final follow up assessment at 1 week
  All the participants in both the groups will be assessed using Patient Global Assessment of Treatment Satisfaction (PGATS) scale.64 65 The question asked will be, ''How satisfied are you overall with the study treatment?'' on a 5-point categorical scale (0 = ''Very dissatisfied''; 1 = ''Dissatisfied''; 2 = ''Neutral or no preference''; 3 = ''Satisfied''; 4 = ''Very satisfied'') at the follow-up assessment point. Mean scores of satisfaction of treatment between the groups will be compared using a t-test.
Difficulty in understanding the information provided by the physiotherapist. | Final follow up assessment at 1 week
  All the participants in both the groups will be asked about the difficulty in understanding the information provided by the physiotherapist. The question asked will be, "How difficult was it for you to understand the information provided by the physiotherapist?" using a on a 5-point Likert Scale, where 1= "Very easy", 2= "Easy", 3= "Neither easy nor difficult", 4= "Difficult", 5= "Very difficult."
Adverse events | Post intervention on day 1, and at final assessment at 1 week.
  All the participants in both the groups will be asked about any adverse events after the treatment. The adverse events will be recorded as a written down verbatim. The type of adverse events will be recorded. The frequency of adverse events in each group will be compared and reported.

SECONDARY OUTCOMES:
Patient-Reported Outcome Measurement Information System (PROMIS) pain interference short form 6b | Baseline assessment and final assessment at 1 week
  5 point, Ordinal scale; It asks respondents to rate how much pain interfered with their daily life (e.g., enjoyment of life, ability to concentrate, day-to-day activities) in past 7 days on 5-point Likert scales (1 = "Not at all," 2 = "A little bit," 3 = "Somewhat," 4 = "Quite a bit," 5 = "Very much"). Total scores can range between 6 to 30. Higher scores indicate more pain interference and worse physical function.
PROMIS pain intensity short form 3b | Baseline assessment and final assessment at 1 week
  5-point, Ordinal scale; It asks the respondents to rate their current pain, worst and average pain intensity in past 7 days on 5-point Likert Scales (1 = "Had no Pain," 2 = "Mild," 3 = "Moderate," 4 = "Severe," and 5 = "Very severe"). Worst pain, average pain, and current pain intensity in the past 7 days are scored on a Likert scale ranging from 1-5. Total score ranges from 3-15, with greater scores indicating more intense pain.
Single-item quality-of-life (QOL) scale | Baseline assessment and final assessment at 1 week
  5-point, Ordinal scale; General quality of life health in the past one week will be assessed on a scale ranging from 0 to 4, by asking the question, "in general, how would you rate your overall quality of life during the past week?" The responses will be recorded on a Likert Scale from 1 = "Poor", 2= "Fair", 3= "Good", 4= "Very good", and 5= "Excellent".2 Greater score indicate better quality of life.
Pain Catastrophizing Scale (PCS) | Baseline assessment and final assessment at 1 week
  A 13 item 5-point, Ordinal scale. Respondents are asked to indicate the degree or frequency with which they have each catastrophizing response listed when they "… are experiencing pain" on a 5-point Likert scale (0 = "Not at all," 1 = "To a slight degree," 2 = "To a moderate degree," 3 = "To a great degree," and 4 = "All the time"). The total PCS score can range from 0 to 52 with higher scores representing higher pain catastrophizing.
Global Rating of Change (GROC) | Final assessment at 1 week
  Single item Score ranges from 1-7, Ordinal scale. Assesses overall improvement since the first assessment. Score ranges from 1 to 7. GROC score =4, indicate no change. Scores greater than 4 indicate greater improvement and scores lower than 4 means greater worsening in health condition.
PROMIS sleep disturbance short form 8b | Baseline assessment and final assessment at 1 week
  5-point, Ordinal scale. It asks respondents to rate sleep related questions on a 5-point Likert scale. Every item is scored on a scale from 1-5. Total scores range from 7 to 35. Greater scores indicate more sleep disturbance.
PROMIS emotional distress- Depression- Short form | Baseline assessment and final assessment at 1 week
  5-point, Ordinal scale. The Depression items asks respondents to indicate the frequency that they have experienced feelings such as worthlessness, helplessness, sadness, hopelessness over the past 7 days on a 5-point verbal rating scale (1 = "Never," 2 = "Rarely," 3 = "Sometimes," 4 = "Often," and 5 = "Always").
10-item Connor Davidson Resilience Scale | Baseline assessment and final assessment at 1 week
  Has 10 items, 4-point, Ordinal scale. Each item is rated by respondents on a 5-point Likert scale: 0 = "Not true at all", 1 = "Rarely true," 2 = "Sometimes true," 3 = "Often true," and 4 = "True nearly all the time". The total score can range from 0 to 40, with higher scores indicating higher resilience.
Use of pain medications and other treatments. | Baseline assessment and final assessment at 1 week
  Names, and dosage of pain medication intake will be recorded. E.g., name of the medicine Dosage in mg Total number of medications taken since the baseline assessment. Other treatments if the patients have undertaken will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Saurab Sharma, MPT, Principal Investigator — Kathmandu University School of Medical Sciences
Locations (1):
- Sahara Physiotherapy Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma S, Jensen MP, Moseley GL, Abbott JH. Results of a feasibility randomised clinical trial on pain education for low back pain in Nepal: the Pain Education in Nepal-Low Back Pain (PEN-LBP) feasibility trial. BMJ Open. 2019 Mar 27;9(3):e026874. doi: 10.1136/bmjopen-2018-026874. PMID 30918037
- [Derived] Sharma S, Jensen MP, Moseley GL, Abbott JH. Pain education for patients with non-specific low back pain in Nepal: protocol of a feasibility randomised clinical trial (PEN-LBP Trial). BMJ Open. 2018 Aug 10;8(8):e022423. doi: 10.1136/bmjopen-2018-022423. PMID 30099402